CLINICAL TRIAL: NCT06441630
Title: A Multicenter, Randomized, Double-blind, Phase III Study to Evaluate the Efficacy and Safety of AD-227A and AD-227B Combination Treatment in Patients with Essential Hypertension
Brief Title: A Study to Evaluate the Efficacy and Safety of Co-administration of AD-227A and AD-227B
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-227P3
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Co-administration of AD-227A and AD-227B (Experimental): AD-227A + AD-227B + Placebo of AD-227C
  Interventions: Drug: AD-227A; Drug: AD-227B; Drug: Placebo of AD-227C
- AD-227A (Active Comparator): AD-227A + Placebo of AD-227B + Placebo of AD-227C
  Interventions: Drug: AD-227A; Drug: Placebo of AD-227B; Drug: Placebo of AD-227C
- Co-administration of AD-227A and AD-227C (Active Comparator): AD-227A + Placebo of AD-227B + AD-227C
  Interventions: Drug: AD-227A; Drug: AD-227C; Drug: Placebo of AD-227B

INTERVENTIONS:
Drug: AD-227A — Per Oral, 1 Tablet, Once a day for 8 weeks
Drug: AD-227B — Per Oral, 1 Tablet, Once a day for 8 weeks
  Arms: Co-administration of AD-227A and AD-227B
Drug: AD-227C — Per Oral, 1 Tablet, Once a day for 8 weeks
  Arms: Co-administration of AD-227A and AD-227C
Drug: Placebo of AD-227B — Per Oral, 1 Tablet, Once a day for 8 weeks
  Arms: AD-227A; Co-administration of AD-227A and AD-227C
Drug: Placebo of AD-227C — Per Oral, 1 Tablet, Once a day for 8 weeks
  Arms: AD-227A; Co-administration of AD-227A and AD-227B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of co-administration of AD-227A and AD-227B in patients with essential hypertension

DETAILED DESCRIPTION:
Essential Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients with Essential Hypertension
* Other inclusions applied

Exclusion Criteria:

* Patient with Secondary Hypertension
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in MSSBP | Baseline to Week8
  Change from Baseline in Mean Sitting Systolic Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Jin Kim, Principal Investigator — Gangnam CHA Medical Center
Locations (1):
- Gangnam CHA Medical Center, Seoul, South Korea